CLINICAL TRIAL: NCT00216528
Title: A Prospective, Open-Label Study to Evaluate Symptomatic Remission in Schizophrenia With Long Acting Risperidone Microspheres (Risperdal Consta)
Brief Title: A Study to Evaluate Symptomatic Remission in Schizophrenia With Long Acting Risperidone Microspheres
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004966
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; risperidone; Intramuscular injection, long-acting risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate symptomatic remission rate in patients with schizophrenia using long acting risperidone microspheres

DETAILED DESCRIPTION:
Although most of Korean schizophrenic patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to daily oral regimen. Long-acting injectable formulation may eliminate this need for daily medication. This is a prospective, open-label, multicenter study to determine the long-term efficacy, especially symptomatic remission rate of long-acting risperidone microspheres administrered in the muscle at 2 week intervals in patients with schizophrenia.

The patients will receive intramuscular injections either 25, 37.5, 50 mg equivalent of risperidone at every 2 weeks for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Subjects with schizophrenia or schizoaffective disorder - Subjects who have experienced relapse or re-admission previously - Subject and/or his/her relative, guardian or legal representative who has signed the informed consent form

Exclusion Criteria:

* First antipsychotic treatment ever - On clozapine during the last 3 months - Serious unstable medical condition, including recent and present clinically relevant laboratory abnormalities - Subjects that are previously on concomitant use of Risperdal Consta within 60 days prior to entry - Previous sensitivity history to risperidone - History or current symptoms of tardive dyskinesia - History of neuroleptic malignant syndrome - Pregnant or breast-feeding female - Female patient of childbearing age without adequate contraception (adequate contraception includes: abstinence, oral contraceptive, intrauterine devices, barrier method (diaphragm or condom) plus spermicide - Norplant TM or Depo-Provera TM. A female patient of childbearing potential must have an adequate contraception and a negative urine pregnancy test at every visit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2005-07; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The symptomatic remission rate at 48 weeks

SECONDARY OUTCOMES:
The change from baseline in Clinical Global Impression-Severity (CGI-S) score at 48 weeks; The change from baseline in SQLS score at 48 weeks; Health-Economic Data

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

REFERENCES:
- [Derived] Lee NY, Kim SH, Cho SJ, Chung YC, Jung IK, Kim CY, Kim DH, Lee DG, Lee YH, Lim WJ, Na YS, Shin SE, Woo JM, Yoon JS, Yoon BH, Ahn YM, Kim YS. A prospective, open-label study to evaluate symptomatic remission in schizophrenia with risperidone long-acting injectable in Korea. Int Clin Psychopharmacol. 2014 Sep;29(5):279-87. doi: 10.1097/YIC.0000000000000030. PMID 24583566